CLINICAL TRIAL: NCT06700668
Title: Active Knee Prosthesis Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts Institute of Technology (Other)
Collaborators: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 0804002682
Record Dates: First submitted 2024-11-04; First posted 2024-11-22 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Transfemoral Amputation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- MIT Powered Knee (Experimental): Subjects wears the MIT powered knee prosthesis.
  Interventions: Device: MIT Powered Knee
- Prescribed prosthesis (No Intervention): Subjects wears their prescribed prosthesis.

INTERVENTIONS:
Device: MIT Powered Knee — MIT powered knee prosthesis developed by the MIT Biomechatronics Group.
  Arms: MIT Powered Knee

SUMMARY:
The purpose of the study is to investigate the clinical and functional outcomes of a powered knee prosthesis for people with a transfemoral amputation in the domain of gait, free space control, and embodiment

ELIGIBILITY:
Inclusion Criteria:

* Male or Female age 22-65.
* The patient must have a unilateral transfemoral amputation .
* The patient must have the ability to ambulate at variable cadence (an expected lower extremity prosthesis functional level of K3 or above).
* The patient must have adequate socket to support the device.

Exclusion Criteria:

* Women who are pregnant.
* Severe co morbidity, atypical skeletal anatomy, or poor general physical/mental health that, in the opinion of the Investigator, will not allow the subject to be a good study candidate (i.e. other disease processes, mental capacity, substance abuse, shortened life expectancy, vulnerable patient population, BMI >40, etc.).

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2008-04-17 (Actual); Primary Completion 2025-07-17 (Actual); Study Completion 2026-07-17 (Estimated)

PRIMARY OUTCOMES:
Metabolic cost | An average of 2 sessions in the span of 1 week
  Effort of participants' walking measured via metabolic cost, which is measured using an mask that measures the Oxygen and Carbon dioxide levels.

SECONDARY OUTCOMES:
Ground reaction force | An average of 2 sessions in the span of 1 week
  Ground reaction forces will be measured via force plates on the ground.
Gait kinematics | An average of 2 sessions in the span of 1 week
  Motion capture data will be collected using a validated system (e.g., Vicon, or similar motion capture software). Reflective markers will be placed on anatomical landmarks following a standard gait model. Kinematic measures, including joint angles (hip, knee, and ankle), step length, stride length, cadence, and walking speed, will be derived.

CONTACTS AND LOCATIONS:
Overall Officials: Hugh Herr, PhD, Principal Investigator — Massachusetts Institute of Technology
Locations (1):
- MIT Media Lab, Cambridge, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided
Subject confidentiality.